CLINICAL TRIAL: NCT04012437
Title: Sphincter Control Training Program Using a App and Electronic Medical Device in the Treatment of Premature Ejaculation: Randomized Controlled Trial
Brief Title: Efficacy of App and Electronic Device in the Treatment of Premature Ejaculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Sexológico Murciano (Other)
Collaborators: Hospital Virgen del Alcazar de Lorca (Unknown)
Responsible Party: Principal Investigator, Jesus Eugenio Rodríguez Martínez, Director of Research Area, Instituto Sexológico Murciano
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISM-SCT-2019-01
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Premature Ejaculation; Masturbation; Medical Device
Keywords: Premature ejaculation; IELT; Medical device
MeSH Terms: conditions — Premature Ejaculation; Masturbation

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Masking Description: A simple blind: The subjects do not know whether they are receiving an experimental treatment or a control treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): .The groups completed Sphincter Control Training over 8 weeks. The SCT consists of 8 different exercises into a mobile app and an educational videos. Its objective is to provide patients with greater knowledge, awareness, and control of the external urethral sphincter. The groups use of a masturbation aid device called Myhixel I from the spanish company New Wellness Concept SL.
  Interventions: Device: Sphincter Control Training (SCT)
- Control (Active Comparator): .The groups completed Sphincter Control Training over 8 weeks. The SCT consists of 8 different exercises into a video tutorial and an educational videos. Its objective is to provide patients with greater knowledge, awareness, and control of the external urethral sphincter.
  Interventions: Behavioral: Sphincter Control Training (SCT)

INTERVENTIONS:
Device: Sphincter Control Training (SCT) — The SCT + device consists of 8 different exercises and an educational session into a app using a masturbation electronic aid device
  Arms: Experimental
Behavioral: Sphincter Control Training (SCT) — The SCT consists of 4 different exercises and an educational session into a app using a masturbation electronic aid device
  Arms: Control

SUMMARY:
Randomized control trial to determine if we can produce increases in the IELT using a new masturbator electronic in subjects with premature ejaculation in combination with a exercise app, producing improvements in the quality and satisfaction of the sexuality of the patient.

DETAILED DESCRIPTION:
This project of research will use one experimental groups, It will manage the affairs the therapy "sphincter control training" (SCT) into app combined with the external device called Myhixel I .Experimental groups will receive therapy with the protocol of exercises SCT.

The main measure will be the "fold increase" (FI) of the IELT, which was calculated using the geometric mean of post-treatment IELTs (period B) divided by the geometric mean of pre-treatment IELTs (period A): FI = (geometric mean of IELT_7wk)/(geometric mean of PRE_IELT)

The efficiency on the EP will see (IELT) reflected in an increase in the times of latency of intravaginal ejaculation and in punctuations of subjective perception, of the therapy on the line base.

The subjects that will be born in mind will be all the interested parties in informing that their answer to the campaign of national advertising that will be started.

The duration of the treatment will be 8 weeks during which a series of exercises app will be practised usin the masturbation device Myhixel I.

The material used in the research will be innocuous and his responsible use does not produce adverse reactions of interest.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years.
* Being in a heterosexual relationship for at least the last 6 months.
* Having a score of >11 on the Premature Ejaculation Diagnostic Tool (PEDT).
* Having a self-reported IELT ≤2 minutes.

Exclusion Criteria:

* A history of alcohol abuse or dependence.
* Having received medication or psychological treatment for PE in the last 6 months.
* Having diabetes.
* The regular use of recreational drugs (except tobacco and caffeine).

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
IELT FOLD INCREASE | 10 weeks
  The main measure will be the "fold increase" (FI) of the IELT, which was calculated using the geometric mean of post-treatment IELTs (period B) divided by the geometric mean of pre-treatment IELTs (period A): FI = (geometric mean of IELT_7wk)/(geometric mean of PRE_IELT)

SECONDARY OUTCOMES:
PEDT | 10 weeks
  The test-retest reliability of the PEDT is .82, and all items discriminate in a statistically significant way between patients with PE and without PE, with a cut-off score for the diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Jesús Rodríguez, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No